CLINICAL TRIAL: NCT04125082
Title: A Single-Site, Investigator-Initiated Study to Evaluate Time in Range in Subjects With Type 2 Diabetes Mellitus Using Mealtime Inhaled Insulin (Afrezza®) Plus Basal Insulin Compared to Multiple Daily Injections
Brief Title: A Study to Evaluate Time in Range in Type 2 Diabetics Using Afrezza® Plus Basal Insulin Compared to Multiple Daily Injections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diabetes and Glandular Disease Clinic (Industry)
Collaborators: Mannkind Corporation (Industry); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-001
Record Dates: First submitted 2019-10-09; First posted 2019-10-14 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Treated With Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Type 2 Diabetics (Other): Participants will be titrated from usual pre-meal insulin plus basal to Afrezza® inhaled insulin plus basal, and will continue on treatment for 14 weeks. Participants will attend study visits at Day 0, Weeks 1, 2, 3, 4, 8, 12 and 16, where insulin titration may be performed based on CGM readings. Participants will receive instruction in carbohydrate counting and corrective insulin dose adjustments.
  Participants will wear CMG throughout the study.
  At final study visit, CGM system will be collected. A1c, FEV1 and Quality of Life Questionnaires will be collected. Pregnancy test will be collected for all females of child-bearing potential. Participants will be transitioned back to Multiple Daily Injections plus basal or may choose to continue on commercial Afrezza® inhaled insulin plus basal
  Interventions: Drug: Afrezza Inhalant Product

INTERVENTIONS:
Drug: Afrezza Inhalant Product — Participants will be titrated from usual pre-meal insulin plus basal to Afrezza® inhaled insulin plus basal, and will continue on treatment for 14 weeks.

SUMMARY:
The purpose of this study is to collect CGM, A1c and Quality of Life data in subjects with Type 2 diabetes before and after transitioning from Multiple Daily Injections to Basal plus Bolus with Afrezza® inhaled insulin. The primary objective is to evaluate the percentage of time spent in goal range without significant hypoglycemia. Additional objectives include evaluation of A1c and Quality of Life data. The expected outcomes are improvement of time in range, no change or improvement in A1c and favorable Quality of Life data

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosed with Type 2 diabetes mellitus treated with multiple daily injections
3. Screening A1c 7.5 % - 11.5% inclusive
4. Willing and able to wear CGM system during the study
5. Willing to use only inhaled insulin (Afrezza®) at meals and for correction
6. Able to understand, speak, read and write English
7. Female of child-bearing potential willing to use contraceptive measures to prevent pregnancy

Exclusion Criteria:

1. Diagnosed with COPD
2. Is an active smoker , or has smoked in the past 6 months
3. Diagnosed with asthma
4. Pregnancy, breast-feeding or planning to become pregnant during study period
5. Have a disease or condition that, in the opinion of the Investigator, could affect subject safety or interfere with their participation in the study
6. Use of oral or injected corticosteroid within 6 weeks of study enrollment
7. Enrollment in another investigational trial at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Time In Range | Week 2 to End of Study
  Evaluation of percentage of time spent in goal range, above (hyperglycemic range) and below (hypoglycemic range) via CGM system from visit week 2 baseline to final study visit with inhaled insulin (Afrezza®).
Hypoglycemia | Week 2 to Week 16
  Incidence of significant hypoglycemic events

SECONDARY OUTCOMES:
Hemoglobin A1c | Week 2 to Week 16
  Evaluation of A1c from visit week 2 baseline to final study visit
Quality of Life Questionnaires | Screening to Week 16
  Evaluation of Diabetes Quality of Life Questionnaires from baseline to final study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kipnes, M.D., Principal Investigator — Diabetes and Glandular Disease Clinic, P.A.
Locations (1):
- Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No